CLINICAL TRIAL: NCT05574803
Title: Using High-definition Transcranial Direct Current Stimulation to Improve Speech Fluency in Cantonese-speaking Adults Who Stutter - A Preliminary Investigation
Brief Title: High-definition tDCS Treatment for Cantonese-speaking Adults Who Stutter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Min Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20210311001
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Stuttering, Adult; Stammering
Keywords: tDCS; Stuttering; Speech therapy; Camperdown Program
MeSH Terms: conditions — Stuttering; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Double-blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): The experimental group will receive 20 minutes of anodal HD-tDCS for five sessions, combined with 20 minutes of behavioural therapy.
  Interventions: Device: Active-tDCS
- Sham tDCS (Sham Comparator): The control group will only receive one minute of anodal HD-tDCS stimulation which aims to create a similar sensation on the scalp as those in the experimental group, with 20 minutes of behavioural therapy.
  Interventions: Device: Sham-tDCS

INTERVENTIONS:
Device: Active-tDCS — Active-tDCS (1 mA) over the supplementary motor area (SMA) for 5 sessions (20 minutes per session, weekly), along with behavioural therapy of speaking tasks (i.e., story narration and conversation) using the minimum prolongation technique based on the Camperdown Program.
  Arms: Active tDCS
Device: Sham-tDCS — Sham-tDCS (1 mA) over the supplementary motor area (SMA) for 5 sessions (one minutes per session, weekly), along with behavioural therapy of speaking tasks (i.e., story narration and conversation) using the minimum prolongation technique based on the Camperdown Program. Participants will receive initial stimulation for one minute, eliciting a tingling sensation on the scalp then it will be discontinued.
  Arms: Sham tDCS

SUMMARY:
The proposed study aims to investigate the effect of combined transcranial direct current stimulation (tDCS) and behavioural speech training in improving speech fluency in Cantonese-speaking adults who stutter (AWS), and to examine its maintenance over a 6-week period.

DETAILED DESCRIPTION:
The proposed study aims to

1. assess the effect of multiple sessions of tDCS over the supplementary motor area (SMA) combined with behavioural speech training on stuttering recovery in terms of a reduction of stuttering severity and increased speech satisfaction in Cantonese-speaking AWS;
2. investigate the maintenance of combined tDCS-behavioural speech training effects on speech fluency and speech satisfaction in Cantonese-speaking AWS over a 6-week period.

Twenty Cantonese-speaking AWS will be randomly assigned to an experimental group and a control group. Both groups will receive behavioral treatment for stuttering, including the speech prolongation technique, for five sessions. Concurrent with behavioural training, the experimental group will receive anodal tDCS (1 mA for 20 minutes), while the control group will receive sham tDCS (1 mA for one minute), over the SMA. Stuttering severity and speech satisfaction will be assessed independently before, immediately after, one week and six weeks after treatment. It is anticipated that AWS will experience reduction in their stuttering severity after stimulation, and the improvement will be maintained for a longer period as compared with receiving behavioural treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated features of stuttering;
* More than 2% of syllables stuttered over three baseline speech samples, as measured by qualified speech therapists.

Exclusion Criteria:

* Personal or family history of epilepsy or seizures
* History of a neurological condition
* Speech disorders
* Hearing impairment
* Metallic foreign body implant
* On medications that lower neural thresholds (e.g. tricyclines, antidepressants, neuroleptic agents, etc.)
* Pregnant
* Had speech therapy for stuttering in the past four months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Stuttering severity [Percent syllables stuttered (%SS)] | Change before, immediately after, one week and six weeks after treatment
  %SS is based on the proportion of spoken syllables that a judge perceives to be stuttered. It will be measured by a qualified speech therapist with prior training in stuttering assessment in Cantonese who will be blinded to the treatment conditions. To establish inter-rater agreement, 20% of the speech samples across different assessment data points will be randomly selected and rated by a second speech therapist.
Stuttering severity [Severity rating (SR)] | Change before, immediately after, one week and six weeks after treatment
  The subjects will be trained to rate their own stuttering severity based on a 9-point SR scale, with 0 = no stuttering, 1 =very mild stuttering, and 8 = the most severe stuttering.

SECONDARY OUTCOMES:
Subject satisfaction | One week and six weeks after treatment
  For the assessment of subject satisfaction regarding the treatment, the following two Likert-type survey questions will be asked:
  1. How much do you think the treatment helped you to speak more fluently? (1 = not at all, 2 = a little, 3 = somewhat, 4 = a lot, 5 = totally); and
  2. How often/much do you think the treatment helped you to feel less stressed in your communication? (1 = never or not at all, 2 = rarely or a little, 3 = sometimes or somewhat, 4 = often or a lot, 5 = always or totally).

CONTACTS AND LOCATIONS:
Overall Officials: Min Ney Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong